CLINICAL TRIAL: NCT00032240
Title: Randomized Trial of a Wedged Insole for Treatment of Osteoarthritis of the Knee
Brief Title: Shoe Inserts for Treating Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P60AR047785 (NIH); P60AR047785 (NIH); NIAMS-076
Record Dates: First submitted 2002-03-12; First posted 2002-03-13 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Biomechanics
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Foot Orthoses

INTERVENTIONS:
Device: Shoe Insert

SUMMARY:
This trial will test shoe inserts for the treatment of knee osteoarthritis, the most common form of knee arthritis. Those with disease on the inner (medial) aspect of the knee will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Medial knee osteoarthritis
* Pain
* No foot problems
* Lives in Boston, Massachusetts Metro area

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2002-02; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T. Felson, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kerrigan DC, Lelas JL, Goggins J, Merriman GJ, Kaplan RJ, Felson DT. Effectiveness of a lateral-wedge insole on knee varus torque in patients with knee osteoarthritis. Arch Phys Med Rehabil. 2002 Jul;83(7):889-93. doi: 10.1053/apmr.2002.33225. PMID 12098144
- [Background] Goggins J, Baker K, Felson D. What WOMAC pain score should make a patient eligible for a trial in knee osteoarthritis? J Rheumatol. 2005 Mar;32(3):540-2. PMID 15742450
- [Derived] Baker K, Goggins J, Xie H, Szumowski K, LaValley M, Hunter DJ, Felson DT. A randomized crossover trial of a wedged insole for treatment of knee osteoarthritis. Arthritis Rheum. 2007 Apr;56(4):1198-203. doi: 10.1002/art.22516. PMID 17393448